CLINICAL TRIAL: NCT03343015
Title: Functional Assessment of the Stomatognathic System, After the Treatment of Edentulous Patients, With Different Methods of Establishing the Centric Relation
Brief Title: Stomatognathic System Assesment, After Different Methods of Establishing the Centric Relation
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Aleksandra Nitecka-Buchta, Principle Investigator DMD PhD, Medical University of Silesia
Other Study IDs: Mandible centralisation
Record Dates: First submitted 2017-10-31; First posted 2017-11-17 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Temporomandibular Disorders
Keywords: TMD, centric relation, complete dentures
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Denture, Complete

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Traditional CR establishing: establishing a CR in traditional way with occlusal wax rims during complete dentures therapy
  Interventions: Procedure: complete dentures
- Gothic arch method: establishing a CR with gothic arch tracing device during complete dentures therapy
  Interventions: Procedure: complete dentures

INTERVENTIONS:
Procedure: complete dentures — therapy with maxilla and mandible dentures

SUMMARY:
Patients with complete dentures were examined after the prosthoddontic treatment with two methods of establishing a centric relation: wax rims and gothic arch tracing method. The effectiveness of establishing a centric relation was evaluated.

DETAILED DESCRIPTION:
In the study subjective experiences of patients, wearing complete dentures, were compared. Two different methods of determining a centric relation were performed: the traditional method using wax occlusal rims and the Gerber method, based on gothic arch tracings. The success rate of establishing a centric relation in both methods was evaluated (rentgenodiagnostics). The influence of the method used to obtain the centric relation on patients stomatognathic system (condyle centralization, pain) was also evaluated. The comparison between two methods was performed and results were analyzed. A centric relation was analyzed in temporomandibular joints and a corelation between TMD symptoms and centric relation was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* TMD according to RDC/TMD group I ,II
* Edentulous patients wearing complete dentures
* Patients agreement for taking part in the study

Exclusion Criteria:

* Analgesic drug addicted patients
* Neurological diseases with headache (migraine, cluster headache)
* Trauma in the head and neck region in the past 2 years

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending dental office in Germany and in Poland, seeking for dental intervention: complete denture
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-02-24 (Actual); Primary Completion 2016-02-20 (Actual); Study Completion 2017-02-20 (Actual)

PRIMARY OUTCOMES:
Mandible condyles centralisation in temporomandibular joints | 1 year
  mandible condylecentral position

SECONDARY OUTCOMES:
Pain intensity changes in Visual Analogue Scale | 1 year
  subjective pain intensity 0-10 points
Anamnestic Index | 1 year
  Evaluation of an anamnestic index according to Helkimo
Dysfunction Index | 1 year
  Evaluation of an dysfunction index

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Baron, Profesor, Study Director — Department of Temporomandibular Disorders and Orthodontics
Locations (1):
- Department of TMD and Orthodontics Silesian Medical University, Zabrze, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Imanimoghaddam M, Madani AS, Mahdavi P, Bagherpour A, Darijani M, Ebrahimnejad H. Evaluation of condylar positions in patients with temporomandibular disorders: A cone-beam computed tomographic study. Imaging Sci Dent. 2016 Jun;46(2):127-31. doi: 10.5624/isd.2016.46.2.127. Epub 2016 Jun 23. PMID 27358820
- [Background] Ammanna S, Rodrigues A, Shetty NS, Shetty K, Augustine D, Patil S. A tomographic study of the mandibular condyle position in partially edentulous population. J Contemp Dent Pract. 2015 Jan 1;16(1):68-73. doi: 10.5005/jp-journals-10024-1637. PMID 25876953
- [Background] Amorim VC, Lagana DC, de Paula Eduardo JV, Zanetti AL. Analysis of the condyle/fossa relationship before and after prosthetic rehabilitation with maxillary complete denture and mandibular removable partial denture. J Prosthet Dent. 2003 May;89(5):508-14. doi: 10.1016/s0022-3913(03)00029-5. PMID 12806330
- [Background] Abdelnabi MH, Swelem AA. Influence of defective complete dentures renewal on TMD; an MRI and clinical controlled prospective study. Gerodontology. 2015 Sep;32(3):211-21. doi: 10.1111/ger.12102. Epub 2013 Dec 16. PMID 24341614
- [Background] Huang M, Hu Y, Yu J, Sun J, Ming Y, Zheng L. Cone-beam computed tomographic evaluation of the temporomandibular joint and dental characteristics of patients with Class II subdivision malocclusion and asymmetry. Korean J Orthod. 2017 Sep;47(5):277-288. doi: 10.4041/kjod.2017.47.5.277. Epub 2017 Jul 27. PMID 28861389
- [Background] Wilkie ND, Hurst TL, Mitchell DL. Radiographic comparisons of condyle-fossa relationships during maxillomandibular registrations made by different methods. J Prosthet Dent. 1974 Nov;32(5):529-33. doi: 10.1016/0022-3913(74)90007-9. No abstract available. PMID 4531485
- [Background] Katzberg RW, Keith DA, Ten Eick WR, Guralnick WC. Internal derangements of the temporomandibular joint: an assessment of condylar position in centric occlusion. J Prosthet Dent. 1983 Feb;49(2):250-4. doi: 10.1016/0022-3913(83)90511-5. PMID 6572265
- [Derived] Nitecka-Buchta A, Proba T, Proba P, Stefanski K, Baron S. Functional Assessment of the Stomatognathic System, after the Treatment of Edentulous Patients, with Different Methods of Establishing the Centric Relation. Pain Res Manag. 2018 Feb 4;2018:1572037. doi: 10.1155/2018/1572037. eCollection 2018. PMID 29623141